CLINICAL TRIAL: NCT00958334
Title: A Multicenter, Open-Label, Safety And Efficacy, Two Year Extension Study of the Selective Progesterone Receptor Modulator Proellex® (CDB-4124) in Pre-Menopausal Women With Symptomatic Leiomyomata Who Have Previously Completed Study ZPU 003
Brief Title: Extension Study of Proellex in Women Who Have Previously Completed Study ZPU 003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZPU-003 Ext
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Proellex 25 mg (Experimental): Two Proellex® 12.5 mg capsules once daily
  Interventions: Drug: Proellex®
- Proellex 12.5 mg (Experimental): One Proellex® 12.5 mg capsules once daily
  Interventions: Drug: Proellex®
- Placebo (Placebo Comparator): Capsule once a day
  Interventions: Drug: Proellex®

INTERVENTIONS:
Drug: Proellex® — 25 mg daily (two 12.5 mg capsules)
  Other Names: CDB-4124; telapristone acetate

SUMMARY:
ZPU-003 EXT is a 2-year extension study of ZPU-003 (NCT00882258) to determine the continued safety and efficacy of Proellex in women who have previously completed the double-blind portion of the study.

DETAILED DESCRIPTION:
ZPU-003 EXT is a 2-year extension study of ZPU-003 (NCT00882258). The purpose of the study is to determine the continued safety and efficacy of Proellex in women who have previously completed the double-blind portion of the study. The desired primary efficacy outcome will be a changes in vaginal bleeding from baseline to 14 months and 17 months on study drug. The total duration of the study is up to 24 months including transition times, off drug intervals, and follow-up visits). It is expected that over a 16 week on drug interval menses will subside and return after a 4-8 week off drug interval (ODI).

ELIGIBILITY:
Inclusion Criteria:

* Completed the ZPU 003 study and met the inclusion/exclusion criteria of that study.

Exclusion Criteria:

* Low or high grade cervical dysplasia, as determined by Papanicolaou (PAP) smear.
* Pregnant or breastfeeding.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2006-09-07 (Actual); Primary Completion 2008-10-15 (Actual); Study Completion 2008-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (11):
- United States (11):
  - Women's Health Research, Phoenix, Arizona
  - Arizona Wellness Centre for Women, Phoenix, Arizona
  - Medical Centre for Clinical Research, San Diego, California
  - Women's Health Care, Inc., San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Insignia Clinical Research (Tampa Bay Women's Center), Tampa, Florida
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - SC Clinical Research Center, Columbia, South Carolina
  - Advances in Health Inc., Houston, Texas
  - Obstetrical & Gynecolgical Associates, PA (OGA), Houston, Texas
  - Women's Clinical Research Centre, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ZPU-003 EXT was an open-label extension study of ZPU-003 (NCT00882258) and all patients received active medication (25 mg of Proellex); results were summarized according to the following groups - subjects who previously received active drug, by dose (12.5 mg and 25 mg) and subjects who previously received placebo in the double-blind ZPU-003 study.
Groups:
- Proellex 25 mg: Participants received Proellex 25 mg by oral administration once per day in NCT00882258. In this extension study participants receive 25 mg Proellex by oral administration of two 12.5 mg capsules. PI discretion to decrease dose to 12.5mg if warranted.
- Proellex 12.5 mg Then 25 mg: Participants received Proellex 12.5 mg. capsule by oral administration once per day in NCT00882258. In this extension study participants receive 25 mg Proellex by oral administration of two 12.5 mg capsules.
- Placebo, Then 25 mg Proellex: Participants received Placebo capsule by oral administration once per day in NCT00882258. In this extension study participants receive 25 mg Proellex by oral administration of two 12.5 mg capsules.
Period: Overall Study
Arm/Group | Proellex 25 mg | Proellex 12.5 mg Then 25 mg | Placebo, Then 25 mg Proellex
Started | 22 | 22 | 21
Completed | 8 | 5 | 8
Not Completed | 14 | 17 | 13

BASELINE CHARACTERISTICS:
Population: Analyses done on ITT Population. ZPU-003 EXT was an open-label extension study of ZPU-003, all patients received active medication (25 mg of Proellex). Results were summarized as follows - subjects who previously received active drug, by dose (12.5 mg and 25 mg) and subjects who previously received placebo in the double-blind ZPU-003 study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Proellex 25 mg | Proellex 12.5 mg Then 25 mg | Placebo, Then 25 mg Proellex | Total
Number analyzed (Participants) | 22 | 22 | 21 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 21 | 65
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (5.55) | 42.6 (5.38) | 40.6 (6.48) | 41.6 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 21 | 65
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: The Change in Menorrhagia From the Baseline of ZPU-003 to the End of Each Off Drug Interval(ODI) Within the ZPU-003 Extension Study and the Baseline of ZPU-003 to the End of ZPU-003 Ext.
Description: An ODI is defined as a time period of less than 3 months during which a return to menses occurs. All statistical endpoints will use the baseline of ZPU-003 Ext for 14-month data and baseline of ZPU-003 for 17-month data.
Time Frame: Baseline to 17 months
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Proellex 25 mg | Proellex 12.5 mg Then 25 mg | Placebo, Then 25 mg Proellex
Number analyzed (Participants) | 22 | 22 | 21
mL
  Baseline | 136.29 (88.12) | 179.95 (119.83) | 130.86 (147.10)
  Change from baseline to end of ODI 1: number analyzed (Participants) | 7 | 7 | 0
  Change from baseline to end of ODI 1 | -41.00 (71.63) | -63.57 (100.83) |
  Change from baseline to end of ODI 2: number analyzed (Participants) | 5 | 6 | 10
  Change from baseline to end of ODI 2 | -38.60 (69.30) | -33.33 (213.63) | -9.90 (125.88)
  Change from baseline to end of ODI 3: number analyzed (Participants) | 5 | 4 | 7
  Change from baseline to end of ODI 3 | -7.00 (69.63) | -222.50 (121.62) | -31.29 (175.46)
  Change from baseline to end of ODI 4: number analyzed (Participants) | 2 | 0 | 0
  Change from baseline to end of ODI 4 | -48.00 (11.31) |  |
  Change from baseline to 17 months: number analyzed (Participants) | 7 | 5 | 8
  Change from baseline to 17 months | 1.43 (94.09) | -211.40 (148.06) | 17.50 (192.88)

2. Secondary Outcome: Change From Baseline of ZPU-003 Ext to 14 Months and 17 Months in Subject's Menstrual Pictogram Scores (mL) (Subjects Evaluable for Menorrhagia Only)
Description: Patient assessed all menstrual products used for bleeding during the month-long time period between study visits. For the total menstrual pictogram score, a lower score indicated less menstrual bleeding, a higher score indicated more menstrual bleeding. Over the course of a menstrual cycle, each pad was scored on an ordinal scale from 1 to 5, each tampon scored either 1, 1.5, 3 or 8, and clots were scored 1, 3 or 5, based on apparent size. Pictogram scored assessments were converted to approximate mL of blood.
Time Frame: Baseline, 14 months, 17 months
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mL of Blood
Arm/Group | Proellex 25 mg | Proellex 12.5 mg Then 25 mg | Placebo, Then 25 mg Proellex
Number analyzed (Participants) | 22 | 22 | 21
mL of Blood
  Change from baseline to month 14: number analyzed (Participants) | 3 | 3 | 1
  Change from baseline to month 14 | -150.67 (66.89) | -248.67 (174.37) | -654.00 (NA) — SD not calculated due to small sample size.
  Change from baseline to month 17: number analyzed (Participants) | 3 | 2 | 0
  Change from baseline to month 17 | -25.33 (48.01) | -230.00 (240.02) |

ADVERSE EVENTS:
Time Frame: 24 months
Description: ZPU-003 EXT was an open-label extension study of ZPU-003 (NCT00882258) and all patients received active medication (25 mg of Proellex); however, results were summarized according to the following groups - subjects who previously received active drug, by dose (12.5 mg and 25 mg) and subjects who previously received placebo in the double-blind ZPU-003 study.
Arm/Group | Proellex 25 mg | Proellex 12.5 mg Then 25 mg | Placebo, Then 25 mg Proellex
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/22 | 1/21
Other Adverse Events (participants affected / at risk) | 19/22 | 18/22 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proellex 25 mg (N=22) | Proellex 12.5 mg Then 25 mg (N=22) | Placebo, Then 25 mg Proellex (N=21)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine Haemorrhage (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Proellex 25 mg (N=22) | Proellex 12.5 mg Then 25 mg (N=22) | Placebo, Then 25 mg Proellex (N=21)
hot flush (General disorders) | 5 | 5 | 8 — Hot flush
headache (Nervous system disorders) | 7 | 2 | 5 — headache, dizziness,carpal tunnel syndrome
nausea (Gastrointestinal disorders) | 2 | 3 | 3
arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
urinary tract infection (Infections and infestations) | 0 | 0 | 5
hepatic enzyme increased (Investigations) | 0 | 1 | 2
joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 1
anxiety (Psychiatric disorders) | 2 | 1 | 0
acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
uterine polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
endometrial thickening (Reproductive system and breast disorders) | 8 | 6 | 2
fatigue (General disorders) | 1 | 1 | 1
dizziness (Nervous system disorders) | 2 | 2 | 0
amenorrhea (Reproductive system and breast disorders) | 5 | 4 | 6
menorrhagia/uterine hemorrhage/metorrhagia (Reproductive system and breast disorders) | 4 | 3 | 2
ovarian cyst (Reproductive system and breast disorders) | 3 | 3 | 1
vulvovaginal mycotic infection (Reproductive system and breast disorders) | 2 | 0 | 2
breast tenderness (Reproductive system and breast disorders) | 3 | 2 | 0
carpal tunnel syndrome (Nervous system disorders) | 2 | 1 | 0
dysmenorrhoea (Reproductive system and breast disorders) | 2 | 1 | 0
breast cyst (Reproductive system and breast disorders) | 1 | 0 | 1
cervical dysplasia (Reproductive system and breast disorders) | 1 | 1 | 0
pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1
vaginitis bacterial (Reproductive system and breast disorders) | 1 | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
diarrhea (Gastrointestinal disorders) | 1 | 1 | 1
vomiting (Gastrointestinal disorders) | 0 | 3 | 0
abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
colitis (Gastrointestinal disorders) | 2 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
influenza (Infections and infestations) | 3 | 1 | 3
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
blood cholesterol increased (Investigations) | 2 | 0 | 0
prothrombin level increased (Investigations) | 1 | 1 | 0
depression (Psychiatric disorders) | 1 | 0 | 1
dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other